CLINICAL TRIAL: NCT03323827
Title: MOLECULAR REGULATION OF MUSCLE GLUCOSE METABOLISM (AIMS 2A, 2B, 3)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Lawrence Mandarino, Professor of Medicine, University of Arizona
Other Study IDs: 1606632714A004
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 2a: Specific Aim 2. To determine how the cytosolic and mitochondrial protein acetylomes are regulated by muscle contraction in insulin sensitive and resistant human volunteers.
  Protocol 2a. Subjects. Two groups (aged 21-65) will be studied: lean (BMI<25), healthy insulin sensitive subjects, and obese (BMI>30) nondiabetics 20 subjects will be enrolled
- Aim 2b: Specific Aim 2. To determine how the cytosolic and mitochondrial protein acetylomes are regulated by muscle contraction in insulin sensitive and resistant human volunteers.
  Protocol 2b (muscle contraction and acetylation) Subjects. Two groups (aged 21-65) will be studied: lean (BMI<25), healthy insulin sensitive subjects, and obese (BMI>30) 32 subjects will be enrolled
- Aim 3: Specific Aim 3. To determine how acetylation of the mitochondrial inner membrane adenine nucleotide translocase ANT1 regulates protein structure and function.
  Subjects. Two groups (aged 21-65) will be studied: lean (BMI<25), healthy insulin sensitive subjects, and obese (BMI>30) 20 subjects will be enrolled.

SUMMARY:
The molecular nature of insulin resistance in human muscle is still incompletely defined. Our data indicate that acetylation of mitochondrial proteins in humans is regulated by muscle contraction and is dysregulated in insulin resistance. Poor function of mitochondria in skeletal muscle is a hallmark of insulin resistance in skeletal muscle. We propose to use a combination of clinical research and mass spectrometry techniques to determine how the cytosolic and mitochondrial protein acetylation is regulated by muscle contraction in insulin sensitive and resistant human volunteers. We will test the hypothesis that mitochondrial protein acetylation is decreased to a greater degree following a bout of exercise in insulin sensitive than in insulin resistant human muscle. Using these techniques we also propose to determine how acetylation of mitochondrial adenine nucleotide translocase (ANT1) at lysines 10, 23, and 92 regulates ANT1 structure and function. Finally, we propose 4) to use a combination of molecular modeling and in vitro assays together with the approach developed in Aim 3 to characterize the role of acetylation in other mitochondrial proteins. Protein targets for this aim will be prioritized based on the potential role of the protein in insulin resistance or mitochondrial function as well as dysregulation of its acetylation state in insulin resistant muscle.

DETAILED DESCRIPTION:
The purpose of this project has been to define the molecular basis for insulin resistance in human muscle. The preceding two cycles of this project were devoted to using proteomics approaches to map and quantify serine/threonine (S/T) phosphorylation sites on insulin receptor substrate (IRS)-1 in skeletal muscle from healthy and insulin resistant humans.

Recent proteomics experiments reveal that another protein modification, lysine acetylation, is more common in non-histone proteins than has been recognized. There are no data, to our knowledge, regarding a relationship between insulin resistance in vivo in human muscle and protein acetylation. We have used proteomics techniques to discover a number of lysine acetylation sites in skeletal muscle proteins in vivo in humans, and this is prominent in mitochondrial proteins. Preliminary data show that mitochondrial protein acetylation is regulated by muscle contraction, and that this response is reduced in insulin resistance. Finally, the mitochondrial inner membrane protein adenine nucleotide translocase (ANT)1 was abundantly acetylated under resting conditions, and its deacetylation in response to contraction was reduced in insulin resistance. Because ANT1 exerts significant physiological control strength for ADP/ATP exchange, and because mitochondrial function is altered in insulin resistance, it is important to characterize this abnormality. Therefore, in order to determine how abnormalities in regulation of lysine acetylation characterize insulin resistant muscle, we propose:

2. To determine how the cytosolic and mitochondrial protein acetylomes are regulated by muscle contraction in insulin sensitive and resistant human volunteers. We will test the hypotheses that:

a. There is differential acetylation of cytosolic or mitochondrial proteins in insulin resistance.

b. Mitochondrial protein acetylation is decreased to a greater degree following a bout of exercise in insulin sensitive than in insulin resistant human muscle.

3. To determine how acetylation of the mitochondrial inner membrane adenine nucleotide translocase ANT1 regulates protein structure and function. We will use mitochondria isolated from human muscle biopsies and molecular dynamics and elastic network modeling to test the hypotheses that:

1. Deacetylation of lysines 10, 23, and 92 increases ANT1 activity.
2. Oxidation of the mitochondrial matrix (increasing the NAD/NADH ratio) raises deacetylation activity and decreases acetylation of ANT1.
3. ANT1 molecular dynamics are altered by acetylation of lysines 10, 23, and 92.

These aims that involve clinical research will be complemented by two aims (Aims 1 and 4) performed entirely in vitro, not using human specimens or data. For context, these aims are listed on page 1 of the accompanying Research Proposal. We have retained the numbering scheme from the original proposal to avoid confusion. Please note that only Aims 2 and 3 involve clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Aim 2a. Subjects. Two groups (aged 21-65) will be studied: lean (BMI<25), healthy insulin sensitive subjects, and obese (BMI>30) nondiabetics 20 subjects will be enrolled

  1. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
  2. Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
  3. Subjects must range in age as described in each specific protocol.
  4. Subjects must have the following laboratory values:

     Hematocrit ≥ 35 vol% Serum creatinine ≤ 1.6 mg/dl AST (SGOT) < 2 times upper limit of normal ALT (SGPT) < 2 times upper limit of normal Alkaline phosphatase < 2 times upper limit of normal Triglycerides < 150 mg/dl. PT 11.7 -14.3 (During Liposyn/heparin infusion, PT will be determined to insure that it is < 1.5-2.0 times the normal value.) PTT 23.0-37.0.

     Aim 2b (muscle contraction and acetylation). Subjects. Two groups (aged 21-65) will be studied: lean (BMI<25), healthy insulin sensitive subjects, and obese (BMI>30) 32 subjects will be enrolled

     Inclusion Criteria
     * Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
     * Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
     * Subjects must range in age as described in each specific protocol.
     * Subjects must have the following laboratory values:

     Hematocrit ≥ 35 vol% Serum creatinine ≤ 1.6 mg/dl AST (SGOT) < 2 times upper limit of normal ALT (SGPT) < 2 times upper limit of normal Alkaline phosphatase < 2 times upper limit of normal Triglycerides < 150 mg/dl. PT 11.7 -14.3 (During Liposyn/heparin infusion, PT will be determined to insure that it is < 1.5-2.0 times the normal value.) PTT 23.0-37.0.

     Aim 3 Subjects. Two groups (aged 21-65) will be studied: lean (BMI<25), healthy insulin sensitive subjects, and obese (BMI>30) 20 subjects will be enrolled.

     Inclusion Criteria
     * Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
     * Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
     * Subjects must range in age as described in each specific protocol.
     * Subjects must have the following laboratory values:

     Hematocrit ≥ 35 vol% Serum creatinine ≤ 1.6 mg/dl AST (SGOT) < 2 times upper limit of normal ALT (SGPT) < 2 times upper limit of normal Alkaline phosphatase < 2 times upper limit of normal Triglycerides < 150 mg/dl. INR < 1.3

     Exclusion Criteria:
* Aim 2a

  * Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded.
  * Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
  * Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>180, diastolic BP>105, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.

Aim 2b Exclusion Criteria

* Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded.
* Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
* Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>180, diastolic BP>105, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.

Aim 3 Exclusion Criteria

* Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded.
* Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
* Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>180, diastolic BP>105, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.
* Healthy controls with BMI less than 25 who have first degree relatives with Type 2 diabetes are at high risk for insulin resistance, this is an exclusion for this study.

Ages: 21 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is described here with respect to the three aims of this project.
  Specific Aim 2. To determine how the cytosolic and mitochondrial protein acetylomes are regulated by muscle contraction in insulin sensitive and resistant human volunteers.
  Aim 2a. Subjects. Two groups (aged 21-65) will be studied: lean (BMI<25), healthy insulin sensitive subjects, and obese (BMI>30) nondiabetics 20 subjects will be enrolled
  Aim 2b (muscle contraction and acetylation). Subjects. Two groups (aged 21-65) will be studied: lean (BMI<25), healthy insulin sensitive subjects, and obese (BMI>30) 32 subjects will be enrolled
  Specific Aim 3. To determine how acetylation of the mitochondrial inner membrane adenine nucleotide translocase ANT1 regulates protein structure and function.
  Subjects. Two groups (aged 21-65) will be studied: lean (BMI<25), healthy insulin sensitive subjects, and obese (BMI>30) 20 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
ANT Acetylation | 2013-2017
  Acetylation of adenine nucleotide translocase 1 at lysine 23 in human muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Mandarino, PHD, Principal Investigator — The University of Arizona
Locations (1):
- The University of Arizona, Tucson, Arizona, United States